CLINICAL TRIAL: NCT06504589
Title: A Research Study to Advance the CF Therapeutics Pipeline for People Without Modulators
Status: Recruiting | Type: Observational
Sponsor: Nicole Hamblett (Other)
Collaborators: Washington University School of Medicine (Other); Florida State University (Other); University of North Carolina, Chapel Hill (Other); University of Toronto (Other); Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor-Investigator, Nicole Hamblett, Professor of Pediatrics, Division of Pulmonary and Sleep Medicine, UW School of Medicine Adjunct Professor, Biostatistics, UW School of Medicine Co-Executive Director, CF Therapeutics Development Network, Seattle Children's Hospital
Organization: Seattle Children's Hospital (Other)
Other Study IDs: REACH-OB-23
Record Dates: First submitted 2024-06-27; First posted 2024-07-17 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Cystic Fibrosis
Keywords: ineligible and/or not taking CFTR modulators; People with CF
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma and white blood cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The REACH study is for people with CF who do not take cystic fibrosis transmembrane conductance regulator (CFTR) modulators. The goal of the REACH study is to collect research data, including health data and specimens, from people with CF who do not take CFTR modulators. This data may be used to inform CF research, help design CF clinical trials and support the development of new treatments for people with CF who do not take CFTR modulators.

Another goal of this study is to learn about research involvement for people with CF who do not take CFTR modulators, engage them in research, and give them an opportunity to learn about what is involved in participating in a CF research study.

DETAILED DESCRIPTION:
People with Cystic Fibrosis (pwCF) who are genetically ineligible and/or not taking cystic fibrosis transmembrane conductance regulator (CFTR) modulators currently face future health that is considerably different from the approximately 90% of pwCF in the United States who benefit from CFTR modulators. New treatments are being advanced for pwCF who are genetically ineligible or not taking CFTR modulators and these therapies will include both nucleic acid-based therapies (NABTs) to address the underlying defect in CFTR and symptomatic therapies aimed at targeting the symptoms of CF. A key concern for this limited and underserved patient population is being able to advance multiple therapeutic programs in parallel. To complete these studies, CF researchers will need to be able to reach this community effectively while also promoting the use of innovative trial designs.

The REACH Study is a prospective, longitudinal, observational research study to obtain research quality (i.e., monitored research) CF outcome data. Primary outcome endpoints of the Core study (collected across all study participants) are aligned with anticipated clinical trial outcome endpoints needed in overall development of therapies for the CF population unable to benefit from CFTR modulators. This study will also include sub-studies to obtain specialized measures which may help inform efficacy and safety evaluations of new therapies by providing CF control data. Finally, this study also seeks to assess research solicitation and research participation for the CF population that is modulator ineligible or not taking modulators. The observational data collected within this study may be used in characterizing this CF population, developing innovative trial designs, for comparison when evaluating new or experimental CF therapies, and/or in CF research.

ELIGIBILITY:
Consent

A. Written informed consent (and assent when applicable) obtained from participant or participant's legal guardian

B. Is willing and able to adhere to the study visit schedule and other protocol requirements

Demographics

A. ≥ 12 years of age at Visit 1

Medical History

A. For persons of child-bearing potential: must not be pregnant at Visit 1 or plan to get pregnant during the 12-month study period

Disease History

A. Documentation of a CF diagnosis as evidenced by one or more clinical features consistent with the CF phenotype and one or more of the following criteria:

* Sweat chloride ≥ 60 mEq/liter by quantitative pilocarpine iontophoresis test (QPIT)
* Two well-characterized disease-causing pathogenic variants in the CFTR gene

or

* One well-characterized disease-causing mutation and a second CFTR variant (with variable or uncharacterized disease-causing potential) and sweat ≥ 30 mmol/liter with permission of the study sponsor-investigators

B. Clinically stable with no significant changes in health status within the 28 days prior to and including Visit 1

C. Does not have a history of lung transplantation

Concomitant Medications

A. Not genetically eligible for a CFTR modulator according to product label indications and/or No use of CFTR modulator for 28 days prior to Visit 1 with no intent to start or restart during the study period

B. No use of an investigational drug within 90 days prior to and including Visit 1

C. Not currently participating in an interventional drug or device trial. Participation in long-term safety follow-up studies (without redosing) and/or behavioral intervention trials is allowed.

D. No initiation of new chronic therapy (e.g., ibuprofen, azithromycin, inhaled tobramycin, Cayston®) within 28 days prior to and including Visit 1

E. No acute use of antibiotics (oral, inhaled or IV) or acute use of systemic corticosteroids for respiratory tract symptoms within 28 days prior to and including Visit 1

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People with CF who are ineligible and/or not taking an approved CFTR modulator and who are not receiving an investigational therapy.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-09-18 (Actual); Primary Completion 2029-08-14 (Estimated); Study Completion 2029-08-14 (Estimated)

PRIMARY OUTCOMES:
Change in ppFEV1 at 12 months | 12 months
  Mean change (standard deviation) in percent predicted forced expiratory volume in 1 second (ppFEV1) as measured by in-clinic spirometry from baseline to 12 months post-baseline.

SECONDARY OUTCOMES:
Change in CFQ-R-RD at 12 months | 12 months
  Mean change (standard deviation) in the Cystic Fibrosis Question - Revised Respiratory Domain (CFQ-R-RD) from Baseline to 12 months post-baseline. Scores for the CFQ-R-RD range from 0 to 100.
Change in home spirometry ppFEV1 at 12 months | 12 months
  Mean change (standard deviation) in percent predicted forced expiratory volume in 1 second (ppFEV1) as measured by home spirometry from baseline to 12 months post-baseline.
Change in LCI 2.5% at 12 months | 12 months
  Mean change (standard deviation) in lung clearance index (LCI) calculated as 1/40th of starting end-tidal concentration of N2 (LCI 2.5%) as measured by multiple breath washout (MBW) from baseline to 12 months post-baseline.
Change in LCI 5% at 12 months | 12 months
  Mean change (standard deviation) in lung clearance index (LCI) calculated as 1/20th of starting end-tidal concentration of N2 (LCI 5%) as measured by multiple breath washout (MBW) from baseline to 12 months post-baseline.
Absolute 12-month change in MCC Index | 12 months
  Mean change (standard deviation) in mucociliary clearance (MCC) index as by the MCC procedure per gamma scintigraphy from baseline to 12 months post-baseline.
Relative 12-month change in MCC Index | 12 months
  Mean change (standard deviation) in mucociliary clearance (MCC) index as by the MCC procedure per gamma scintigraphy from baseline to 12 months post-baseline divided by the baseline MCC index.

CONTACTS AND LOCATIONS:
Overall Officials: Deepika Polineni, MD, MPH, Principal Investigator — Washington University School of Medicine; Nicole Mayer-Hamblett, PhD, Principal Investigator — Seattle Children's Hospital; Scott Donaldson, MD, Principal Investigator — University of North Carolina, Chapel Hill; Felix Ratjen, MD, Principal Investigator — University of Toronto
Locations (68):
- United States (68):
  - The Children's Hospital Alabama, University of Alabama at Birmingham, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Tucson Cystic Fibrosis Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of California San Diego, La Jolla, California
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Stanford University Medical Center, Palo Alto, California
  - University of California, San Francisco - Adult Center, San Francisco, California
  - University of California, San Francisco - Peds Center, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - National Jewish Health, Denver, Colorado
  - University of Florida, Gainesville, Florida
  - University of Miami, Miami, Florida
  - Central Florida Pulmonary Group, Orlando, Florida
  - Tampa General Hospital, Tampa, Florida
  - Children's Healthcare of Atlanta and Emory University, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - Saint Luke's Cystic Fibrosis Center of Idaho, Boise, Idaho
  - Northwestern University, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Tulane University, Metairie, Louisiana
  - John Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Massachusetts Memorial Health Care, Worcester, Massachusetts
  - University of Michigan, Michigan Medicine, Ann Arbor, Michigan
  - Wayne State University Harper University Hospital, Detroit, Michigan
  - Corewell Health Helen DeVos, Grand Rapids, Michigan
  - The Minnesota Cystic Fibrosis Center, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Billings Clinic, Billings, Montana
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Morristown Medical Center, Morristown, New Jersey
  - The Cystic Fibrosis Center of Western New York, Buffalo, New York
  - Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Columbia University Cystic Fibrosis Program, New York, New York
  - University of Rochester Medical Center Strong Memorial, Rochester, New York
  - New York Medical College at Westchester Medical Center, Valhalla, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital/University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cystic Fibrosis Program, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - Oregon Health & Sciences University, Portland, Oregon
  - Hershey Medical Center Pennsylvania State University, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Children's Hospital - Midlands, Columbia, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - University of Texas Southwestern / Children's Health, Dallas, Texas
  - University of Texas Southwestern, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - Adult Cystic Fibrosis Center at the University of Utah, Salt Lake City, Utah
  - Inova L.J. Murphy Pediatric CF Program, Fairfax, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Providence Medical Group, Cystic Fibrosis Clinic, Spokane, Washington
  - West Virginia University - Morgantown, Morgantown, West Virginia
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No